CLINICAL TRIAL: NCT02026193
Title: IVF Hyper-responders: Oocyte Vitrification Compared With Embryo Freezing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Shahar Kol MD, Director, IVF Unit, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMB-0439-13
Record Dates: First submitted 2013-12-30; First posted 2014-01-01 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oocyte vitrification (Experimental): All retrieved mature oocytes will be vitrified.
  Interventions: Procedure: oocyte vitrification
- embryo freezing (Active Comparator): All retrieved oocytes will be fertilized, and resulting embryos will be frozen.
  Interventions: Procedure: embryo freezing

INTERVENTIONS:
Procedure: oocyte vitrification
  Arms: oocyte vitrification
Procedure: embryo freezing
  Arms: embryo freezing

SUMMARY:
The chances to achieve pregnancy after retrieving >15 oocytes are not good, probably because of bad effect on the endometrium (uterine inner lining). Therefore, in most such cases the investigators prefer to freeze all embryos, and transfer in a thaw cycle. With the introduction of oocyte vitrification (very fast cooling) technology, a new option emerged: to freeze un-fertilized eggs, to be fertilized and used later in a thaw cycle.

The purpose of this study is to compare the outcome of these two approaches.

ELIGIBILITY:
Inclusion Criteria:

* IVF patients
* ovulation trigger with Decapeptyl 0.2 mg because of ovarian hyper-response: E2 on trigger day .12,000 pmol/l and/or >15 oocytes.
* Normal uterus

Exclusion Criteria:

* <20% fertilization rate

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- IVF Unit, Rambam medical Center, Haifa, Israel, Israel

REFERENCES:
- [Background] Devroey P, Polyzos NP, Blockeel C. An OHSS-Free Clinic by segmentation of IVF treatment. Hum Reprod. 2011 Oct;26(10):2593-7. doi: 10.1093/humrep/der251. Epub 2011 Aug 9. PMID 21828116

RESULTS

PARTICIPANT FLOW:
Groups:
- Oocyte Vitrification: All retrieved mature oocytes will be vitrified.
  oocyte vitrification
- Embryo Freezing: All retrieved oocytes will be fertilized, and resulting embryos will be frozen.
  embryo freezing
Period: Overall Study
Arm/Group | Oocyte Vitrification | Embryo Freezing
Started | 3 | 8
Completed | 3 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oocyte Vitrification | Embryo Freezing | Total
Number analyzed (Participants) | 3 | 8 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 8 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (5.5) | 25 (2.6) | 28.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 3 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Fetal Heart Activity 1 Month Post Embryo Transfer
Description: Fetal heart activity as demonsrated by vaginal ultrasound 1 month post embryo transfer
Time Frame: 1 month after embryo transfer
Measure: Number; unit: participants with fetal heart activity
Arm/Group | Oocyte Vitrification | Embryo Freezing
Number analyzed (Participants) | 3 | 8
participants with fetal heart activity | 0 | 4

ADVERSE EVENTS:
Arm/Group | Oocyte Vitrification | Embryo Freezing
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/8
Other Adverse Events (participants affected / at risk) | 0/3 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No